CLINICAL TRIAL: NCT01276158
Title: Ultrasound-image Versus Doppler-guided Radial Artery Cannulation in Infants and Small Children
Brief Title: Pediatric Radial Arterial Cannulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Kenichi Ueda, Clinical Associate Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200905711
Record Dates: First submitted 2011-01-11; First posted 2011-01-13 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultrasound (Active Comparator): Arterial line placed with Ultrasound guidance.
  Interventions: Procedure: Ultrasound
- Doppler (Active Comparator): Arterial line placed with doppler guidance
  Interventions: Procedure: Doppler

INTERVENTIONS:
Procedure: Ultrasound — Ultrasound used to place arterial line
  Arms: Ultrasound
Procedure: Doppler — Doppler used to place arterial line
  Arms: Doppler

SUMMARY:
This prospective randomized study was designed to compare ultrasound guided technique with Doppler assisted technique for radial arterial cannulation in infant and small children.

DETAILED DESCRIPTION:
In infants, percutaneous cannulation of radial artery requires considerable expertise. People have been using Doppler guided radial artery cannulation technique to improve success rate for more than 20 years. Recently, Ultrasound sonography has been utilized for central line placement in pediatrics. The purpose of this study is whether ultrasound guided radial artery cannulation technique improves the success rate compared to traditional doppler guided technique.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria

  1. Pediatric patient undergoing scheduled major surgery which require continuous arterial pressure monitoring
  2. Term neonates and children < 4 years old weighing >/= 3 kg and < 12 kg

Exclusion Criteria:

* Exclusion criteria

  1. Patients with a skin wound or infection around puncture site
  2. Abnormal circulation in the hand (known vascular compromise, mottling, cool skin temp relative to other hand, poor capillary refill)
  3. Recent radial arterial puncture (less than 1 month)
  4. Any emergency surgery or profound hemodynamic instability requiring urgent arterial cannulation.

Max Age: 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The primary object is to compare the first attempt success rate between each group. | 10 minutes

SECONDARY OUTCOMES:
As a secondary object, a comparison will be made between groups for overall Success rate within a 10 minute time period. | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Ueda, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No